CLINICAL TRIAL: NCT02019901
Title: A Randomized, Controlled Study Evaluating the Efficacy of Person-centered, Tight Control Nurse-led Clinic of Patients With Established Rheumatoid Arthritis and Moderate to High Disease Activity Compared to Patients Receiving Regular Care
Brief Title: GotNet Study, The Gothenburg Nurse-led Tight Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Ulrika Bergsten, RN, PHD, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GotNet 2014 SU
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Person-centered care; Tight control
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Practice Patterns, Nurses'

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular care (No Intervention): The control-group is treated according to "care as usual" with visits to physician every 6th month.
- Nurse-led clinic (Experimental): Nurse-led visits every 6th week, with structured person-centered care and evaluation of disease activity. If disease remission is not reached, pharmacological treatment including both short-term (intra-articular and oral steroids) and long-term alterations (DMARDs and biologics) is modified according to a predefined algorithm.
  Interventions: Other: Nurse-led clinic

INTERVENTIONS:
Other: Nurse-led clinic
  Arms: Nurse-led clinic

SUMMARY:
Purpose: To compare a nurse-led clinic including person-centered care and tight control with "care as usual" in patients with rheumatoid arthritis (RA) and moderate/ high disease activity.

Project description: Study population: Patients with RA, 18-80 yrs old, with moderate/ high Disease Activity Score of 28 joints (DAS28 > 3.8) and disease duration > 2 yrs in a 6-month randomized controlled study with a 6 month open follow-up. Intervention group (N=60): Nurse-led visits every 6th week, with structured person-centered care and evaluation of disease activity. If disease remission is not reached, pharmacological treatment including both short-term (intra-articular and oral steroids) and long-term alterations (DMARDs and biologics) is modified according to a predefined algorithm. The control group (N=60) is treated according to "care as usual" with visits to physician every 6th month. Outcome measures: Primary outcome measure is change in Diseases Activity Score (DAS). Secondary outcomes are quality of life, self-efficacy, disability, emotional well-being, pain, fatigue, sleep and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and <80 years of age
* Signed and dated informed consent form before the start of any specific protocol procedures
* Fulfill the 1987 ACR criteria or the 2010 ACR/EULAR criteria for RA with disease duration of >2 years
* Moderate to high disease activity (DAS28 >3.8)
* ≥2 swollen joints

Exclusion Criteria:

* Diagnosis of any other inflammatory arthritis
* History of chronic infection, recent serious or life-threatening infection within 6 months
* Concurrent malignancy, a history of malignancy or current or recent history of severe, progressive, and/or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological or cerebral disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Change in Disease activity score (DAS28) | Baseline, week 26 and 50
  The primary outcome constitute of DAS28, an index comprising the number of tender and swollen joints, patients global health assessment and erythrocyte sedimentation rate

SECONDARY OUTCOMES:
Proportion of patients with low Disease activity score (DAS28) | Baseline, week 26 and 50
Proportion of patients with remisson according to Disease activity score (DAS28) | Baseline, week 26 and 50
Health assessment questionnaire (HAQ) | Baseline, week 26 and 50
  Measures functional status
EuroQol (EQ-5D) | Baseline, week 26 and 50
  Measures health status, allowing computation of cost-effectiveness
Visual analogue scale for pain (VAS-pain) | Baseline, week 26 and 50
  Measures the patient's pain
Visual analogue scale fatigue (VAS-Fatigue) | Baseline, week 26 and 50
  Measures the patient's fatigue.
Visual analogue scale general health (VAS-general health) | Baseline, week 26 and 50
  Measures the patient's general health.
Effective Consumer Survey 17 (EC17) | Baseline, week 26 and 50
  Measures patients' perception of their knowledge, attitudes and behaviors about self-management skills
Rheumatoid Arthritis Impact of Disease (RAID) score, | Baseline, week 26 and 50
  A patient-derived composite measure of the impact of the disease
The beliefs about medicines questionnaire (BMQ) | Baseline,week 26 and 50
  Assessing patients' perceptions and expectation about medicines
Numerical Rating Scale (NRS) about satisfaction with care | Baseline, week 26 and 50
  Measures satisfaction with rheumatology care

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Jacobsson, Professor, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Bergsten U, Almehed K, Baigi A, Jacobsson LTH. A randomized study comparing regular care with a nurse-led clinic based on tight disease activity control and person-centred care in patients with rheumatoid arthritis with moderate/high disease activity: A 6-month evaluation. Musculoskeletal Care. 2019 Sep;17(3):215-225. doi: 10.1002/msc.1403. Epub 2019 Jun 20. PMID 31219668